CLINICAL TRIAL: NCT02889224
Title: In Vivo Study of Interactions Between the Endocannabinoid System and the Corticotropic Axis in Man
Acronym: VISECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2010/34
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cushing's Syndrome
Keywords: Obesity; Cortisol; Hydrocortisone; Endocannabinoïds
MeSH Terms: conditions — Cushing Syndrome; Obesity | interventions — Adiposity; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese (Active Comparator): Subjects with BMI between 30 - 40 kg/m2 and no alteration of corticotrope axis.
  Interventions: Other: Obese
- Hypercortisolism (Experimental): Subject with BMI between 18 - 40 kg/m2 and presenting a hypercortisolism defined by HAS (Haute Autorité de Santé).
  Interventions: Procedure: Hypercortisolism
- Hydrocortisone (Experimental): Subject with BMI between 18 - 30 kg/m2 and with adrenal or corticotrope failure
  Interventions: Other: Hydrocortisone
- Control (Experimental): Subject with BMI between 18 - 30 kg/m2 and with a pituitary or adrenal tumor without effect on corticotrope axis.
  Interventions: Other: Control

INTERVENTIONS:
Other: Obese
  Arms: Obese
Procedure: Hypercortisolism
  Arms: Hypercortisolism
Other: Hydrocortisone
  Arms: Hydrocortisone
Other: Control
  Arms: Control

SUMMARY:
Working hypothesis: the interactions between the endogenous endocannabinoïds (ECS) - and cortisol, the end product of the Hypothalamo-Pituitary-Adrenal (HPA) axis may play a role in the pathophysiology of Cushing's syndrome.

The investigators speculate that:

* acute or chronic variations in plasma cortisol may induce changes in the activity of the ECS
* that there is a circadian rhythm of the ECS driven by the rythm of plasma cortisol

DETAILED DESCRIPTION:
The study aim to identify the relationship between the ECS and the HPA axis in humans with a main objective to assess if Cushing's syndrome induces changes in the ECS activity.

For this purpose:

1. the investigors will compare plasma levels of ECS between obese controls and patients with Cushing's syndrome
2. the investigors will compare plasma levels of ECS in patients with Cushing's syndrome before and immediately after curative surgery
3. the investigors will compare plasma levels of ECS in patients with hypoadrenalism before and after the intake of substitutive doses of hydrocortisone
4. the investigors will evaluate the plasma levels of ECS during a short synacthen test in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

For all patients groups:

* Age ≥ 18,
* Social security.

" Hypercortisolism " group:

* 18 < BMI < 40 kg/m2,
* Cushing's syndrome in front of :
* impaired 1 mg dexamethasone test (08:00 A.M. cortisol > 50 nmol/L)
* qualitative and quantitative disrupted circadian rhythm of cortisol with increased plasma concentrations
* free urinary cortisol upper normal range (90 µg/24H),
* Hypercortisolism that can be treated with surgery (adrenal adenoma treated with adrenalectomy or Cushing disease treated with pituitary surgery).

" Obese " group:

* Obese patients: 30 < BMI < 40 kg/m2,
* Normal HPA axis function:
* 08:00 A.M. cortisol > 250 nmol/L and peak above 550 nmol/L after 1 mg SST,
* Normal 24H free urinary cortisol and dexamethasone test. " Control " group:
* Lean or overweight patients (18 < BMI < 30 kg/m2),
* Non cortisol secreting pituitary or adrenal tumor,
* Patient in whom a biological evaluation of the HPA axis is recommended.

" Hydrocortisone " group:

* Lean or overweight patients (18 < BMI < 30 kg/m2),
* Primary or secondary adrenal insufficiency,
* With a need for hydrocortisone supplementation.

Exclusion Criteria:

* Patients with eating disorders, major depressive disorders or psychiatric disorders other than Cushing's syndrome,
* Cannabis consumption, alcoholism or drug addiction,
* Active smoking,
* cortisone treatment other than hydrocortisone,
* Pregnancy or feeding,
* Surgery for obesity,
* Incapability,
* Pathology that is life-threatening in the short term,
* Any situation that interfere with study or is risked for patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Fluctuations of 2-AG (2-arachidonoyl-Glycérol) plasma concentration in relationship to cortisol plasma concentration in obese arm compare to hypercortisolism arm. | Baseline
  The primary outcome will be assessed by a measurement of plasma concentration of 2-AG during the circadian rhythm of ACTH/cortisol.

SECONDARY OUTCOMES:
Measurement of plasma concentration of AEA (Anandamide), OEA (Oleoyl-EthanolAmide) and PEA (Palmitoyl-EthanolAmide) endocannabinoïds associated with variations of plasma cortisol in hypercortisolism arm | Baseline and day 6
  The secondary outcome wille be assessed by a measurement of plasma concentration of AEA, OEA and PEA during the circadian rhythm of ACTH/cortisol.
Measurement of plasma concentration of AEA (Anandamide), OEA (Oleoyl-EthanolAmide) and PEA (Palmitoyl-EthanolAmide) endocannabinoïds associated with variations of plasma cortisol in hydrocortisone arm | Baseline
  Measurement of plasma concentration of AEA, OEA and PEA on 07:30 A.M. ± 1 hour (fasting), 08:00 A.M. ± 1 hour (fasting), 09:00 A.M. ± 1 hour, 10:00 A.M. ± 1 hour, 04:00 P.M. ± 1 hour
Measurement of plasma concentration of AEA (Anandamide), OEA (Oleoyl-EthanolAmide) and PEA (Palmitoyl-EthanolAmide) endocannabinoïds in control arm who have no cortisol production problem. | Baseline
  Measurement of plasma concentration of AEA, OEA and PEA during the circadian rhythm of ACTH/cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service d'Endocrinologie, Hopital Haut-Leveque, Pessac, France

IPD SHARING:
Plan to Share IPD: No